CLINICAL TRIAL: NCT00622284
Title: A Randomised Double-blind, Active-controlled Parallel Group Efficacy and Safety Study of BI 1356 ( 5.0 mg, Administered Orally Once Daily) Compared to Glimepiride Over Two Years in Type 2 Diabetic Patients With Insufficient Glycaemic Control Despite Metformin Therapy
Brief Title: Efficacy and Safety of BI 1356 in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.20; 2007-004585-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

ARMS (2):
- BI 1356 5mg, once daily (Experimental): patient to receive a tablet containing 5mg BI 1356 plus one (two in US) inactive placebo capsule matching Glimepiride
  Interventions: Drug: Placebo identical to Glimepiride 1mg or 2mg or 3mg or 4 mg; Drug: BI 1356
- Glimepiride (Active Comparator): patient to receive 1mg or 2mg or 3mg (not in US) or 4mg Glimepiride capsule plus one inactive placebo tablet matching BI 1356 (plus one inactive placebo capsule in US)
  Interventions: Drug: Placebo identical to BI 1356 5mg; Drug: Glimepiride

INTERVENTIONS:
Drug: Placebo identical to BI 1356 5mg — Placebo tablet once daily
  Arms: Glimepiride
Drug: Placebo identical to Glimepiride 1mg or 2mg or 3mg or 4 mg — Placebo tablets once daily
  Arms: BI 1356 5mg, once daily
Drug: BI 1356 — 5mg, once daily in the morning for 104 weeks
  Arms: BI 1356 5mg, once daily
Drug: Glimepiride — 1mg or 2mg or 3mg or 4mg in the morning for 104 weeks
  Arms: Glimepiride

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 1356 (5.0 mg daily) compared to glimepiride given for 104 weeks as add-on therapy to preferably > 1500 mg metformin in patients with type 2 diabetes mellitus with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with a diagnosis of type 2 diabetes mellitus and previously treated with metformin alone or with metformin and one other oral antidiabetic drug
2. Glycosylated haemoglobin (HbA1c) 6.0 - 9.0% at screening for patients treated with metformin and one other oral antidiabetic drug
3. HbA1c 6.5 - 10.0% at screening for patients treated with metformin alone
4. HbA1c 6.5 - 10.0% at beginning of the placebo run-in phase

Exclusion criteria:

1. Myocardial infarction, stroke or transient ischemic attack (TIA)
2. Impaired hepatic function
3. Renal failure or renal impairment
4. Treatment with rosiglitazone or pioglitazone within 6 months prior to screening
5. Treatment with insulin or glucagon-like peptide 1 (GLP-1) analogue/antagonists within 3 months prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (221):
- United States (23):
  - 1218.20.10033 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1218.20.10003 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.20.10020 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.20.10035 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.20.10037 Boehringer Ingelheim Investigational Site, Los Gatos, California
  - 1218.20.10034 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 1218.20.10023 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1218.20.10030 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 1218.20.10028 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1218.20.10006 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1218.20.10022 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 1218.20.10032 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1218.20.10031 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1218.20.10013 Boehringer Ingelheim Investigational Site, Mentor, Ohio
  - 1218.20.10045 Boehringer Ingelheim Investigational Site, Perrysburg, Ohio
  - 1218.20.10042 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1218.20.10024 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.20.10002 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.20.10007 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.20.10036 Boehringer Ingelheim Investigational Site, Murray, Utah
  - 1218.20.10029 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1218.20.10009 Boehringer Ingelheim Investigational Site, Federal Way, Washington
  - 1218.20.10026 Boehringer Ingelheim Investigational Site, Renton, Washington
- Bulgaria (5):
  - 1218.20.35201 Boehringer Ingelheim Investigational Site, Sofia
  - 1218.20.35202 Boehringer Ingelheim Investigational Site, Sofia
  - 1218.20.35203 Boehringer Ingelheim Investigational Site, Sofia
  - 1218.20.35207 Boehringer Ingelheim Investigational Site, Sofia
  - 1218.20.35204 Boehringer Ingelheim Investigational Site, Stara Zagora
- Denmark (7):
  - 1218.20.45006 Boehringer Ingelheim Investigational Site, Aalborg
  - 1218.20.45001 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1218.20.45011 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1218.20.45013 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1218.20.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1218.20.45003 Boehringer Ingelheim Investigational Site, København NV
  - 1218.20.45007 Boehringer Ingelheim Investigational Site, Odense
- France (74):
  - 1218.20.3307A Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307B Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307C Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307D Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307E Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307F Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307G Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307H Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3307I Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3310A Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3310B Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3310C Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3310D Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3310E Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3312A Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3312B Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3312C Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3312D Boehringer Ingelheim Investigational Site, Joué Les Tours Cedex
  - 1218.20.3308A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3308C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3308D Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3308E Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3308F Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3309A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3309B Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3309C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3309D Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3309E Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3311A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3311B Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3311C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3313A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3313B Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3313C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3313D Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314B Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314D Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314E Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3314F Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.20.3301A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302C Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302D Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302E Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302G Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302H Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3302I Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303B Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303C Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303D Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303E Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303G Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303H Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3303I Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304B Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304C Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304D Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304F Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3304H Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3305A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3305B Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3305H Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306B Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306D Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306F Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306G Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306H Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3306I Boehringer Ingelheim Investigational Site, Nantes
  - 1218.20.3311D Boehringer Ingelheim Investigational Site, Potigny
- Germany (28):
  - 1218.20.49004 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1218.20.49028 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 1218.20.49022 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.20.49024 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1218.20.49012 Boehringer Ingelheim Investigational Site, Cologne
  - 1218.20.49020 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.20.49018 Boehringer Ingelheim Investigational Site, Flörsheim
  - 1218.20.49015 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1218.20.49006 Boehringer Ingelheim Investigational Site, Großheirath
  - 1218.20.49025 Boehringer Ingelheim Investigational Site, Haag
  - 1218.20.49016 Boehringer Ingelheim Investigational Site, Hamburg
  - 1218.20.49029 Boehringer Ingelheim Investigational Site, Hanover
  - 1218.20.49021 Boehringer Ingelheim Investigational Site, Hatten
  - 1218.20.49017 Boehringer Ingelheim Investigational Site, Kelkheim
  - 1218.20.49005 Boehringer Ingelheim Investigational Site, Künzing
  - 1218.20.49010 Boehringer Ingelheim Investigational Site, Leipzig
  - 1218.20.49003 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.20.49007 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1218.20.49008 Boehringer Ingelheim Investigational Site, Rednitzhembach
  - 1218.20.49027 Boehringer Ingelheim Investigational Site, Saaldorf
  - 1218.20.49014 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1218.20.49019 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1218.20.49030 Boehringer Ingelheim Investigational Site, Speyer
  - 1218.20.49002 Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
  - 1218.20.49009 Boehringer Ingelheim Investigational Site, Unterschneidheim
  - 1218.20.49026 Boehringer Ingelheim Investigational Site, Wangen
  - 1218.20.49011 Boehringer Ingelheim Investigational Site, Westerkappeln
  - 1218.20.49013 Boehringer Ingelheim Investigational Site, Würzburg
- Hong Kong (3):
  - 1218.20.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1218.20.85202 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1218.20.85204 Boehringer Ingelheim Investigational Site, Hong Kong
- Hungary (8):
  - 1218.20.36208 Boehringer Ingelheim Investigational Site, Ajka
  - 1218.20.36205 Boehringer Ingelheim Investigational Site, Baja
  - 1218.20.36204 Boehringer Ingelheim Investigational Site, Békéscsaba
  - 1218.20.36206 Boehringer Ingelheim Investigational Site, Hódmezövásárhely
  - 1218.20.36202 Boehringer Ingelheim Investigational Site, Makó
  - 1218.20.36201 Boehringer Ingelheim Investigational Site, Miskolc
  - 1218.20.36207 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 1218.20.36203 Boehringer Ingelheim Investigational Site, Szentes
- India (8):
  - 1218.20.91022 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.20.91024 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1218.20.91025 Boehringer Ingelheim Investigational Site, Gujarat
  - 1218.20.91023 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1218.20.91021 Boehringer Ingelheim Investigational Site, Kochi
  - 1218.20.91020 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.20.91027 Boehringer Ingelheim Investigational Site, Patna
  - 1218.20.91026 Boehringer Ingelheim Investigational Site, Tamilnadu
- Ireland (6):
  - 1218.20.35307 Boehringer Ingelheim Investigational Site, Co. Cork
  - 1218.20.35304 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 1218.20.35306 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 1218.20.35310 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 1218.20.35308 Boehringer Ingelheim Investigational Site, Dublin
  - 1218.20.35303 Boehringer Ingelheim Investigational Site, Waterford
- Italy (10):
  - 1218.20.39034 Boehringer Ingelheim Investigational Site, Catania
  - 1218.20.39027 Boehringer Ingelheim Investigational Site, Chieti
  - 1218.20.39029 Boehringer Ingelheim Investigational Site, Codogno (lo)
  - 1218.20.39021 Boehringer Ingelheim Investigational Site, Genova
  - 1218.20.39033 Boehringer Ingelheim Investigational Site, Perugia
  - 1218.20.39022 Boehringer Ingelheim Investigational Site, Pordenone
  - 1218.20.39028 Boehringer Ingelheim Investigational Site, Ravenna
  - 1218.20.39030 Boehringer Ingelheim Investigational Site, Roma
  - 1218.20.39032 Boehringer Ingelheim Investigational Site, Roma
  - 1218.20.39020 Boehringer Ingelheim Investigational Site, Siena
- Netherlands (9):
  - 1218.20.31023 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.20.31014 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1218.20.31016 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1218.20.31011 Boehringer Ingelheim Investigational Site, Ewijk
  - 1218.20.31018 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 1218.20.31012 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1218.20.31022 Boehringer Ingelheim Investigational Site, Rilland
  - 1218.20.31019 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1218.20.31013 Boehringer Ingelheim Investigational Site, Wildervank
- Norway (5):
  - 1218.20.47005 Boehringer Ingelheim Investigational Site, Fevik
  - 1218.20.47004 Boehringer Ingelheim Investigational Site, Fornebu
  - 1218.20.47002 Boehringer Ingelheim Investigational Site, Hamar
  - 1218.20.47001 Boehringer Ingelheim Investigational Site, Rud
  - 1218.20.47003 Boehringer Ingelheim Investigational Site, Sandvika
- Poland (9):
  - 1218.20.48210 Boehringer Ingelheim Investigational Site, Bialystok
  - 1218.20.48208 Boehringer Ingelheim Investigational Site, Gdynia
  - 1218.20.48207 Boehringer Ingelheim Investigational Site, Krakow
  - 1218.20.48201 Boehringer Ingelheim Investigational Site, Lodz
  - 1218.20.48202 Boehringer Ingelheim Investigational Site, Lodz
  - 1218.20.48203 Boehringer Ingelheim Investigational Site, Olsztyn
  - 1218.20.48206 Boehringer Ingelheim Investigational Site, Torun
  - 1218.20.48205 Boehringer Ingelheim Investigational Site, Warsaw
  - 1218.20.48209 Boehringer Ingelheim Investigational Site, Warsaw
- South Africa (6):
  - 1218.20.27007 Boehringer Ingelheim Investigational Site, Bellville
  - 1218.20.27002 Boehringer Ingelheim Investigational Site, Cape Town
  - 1218.20.27006 Boehringer Ingelheim Investigational Site, Durban
  - 1218.20.27004 Boehringer Ingelheim Investigational Site, Lenasia
  - 1218.20.27005 Boehringer Ingelheim Investigational Site, Lenasia
  - 1218.20.27003 Boehringer Ingelheim Investigational Site, Pretoria
- Sweden (4):
  - 1218.20.46003 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.20.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.20.46002 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.20.46004 Boehringer Ingelheim Investigational Site, Uppsala
- United Kingdom (16):
  - 1218.20.44108 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 1218.20.44115 Boehringer Ingelheim Investigational Site, Blackpool
  - 1218.20.44110 Boehringer Ingelheim Investigational Site, Bradford-on-Avon
  - 1218.20.44102 Boehringer Ingelheim Investigational Site, Buckshaw Village, Chorley
  - 1218.20.44114 Boehringer Ingelheim Investigational Site, Cheadle
  - 1218.20.44116 Boehringer Ingelheim Investigational Site, Chestfield, Whitstable
  - 1218.20.44109 Boehringer Ingelheim Investigational Site, Chippenham
  - 1218.20.44113 Boehringer Ingelheim Investigational Site, Dundee
  - 1218.20.44105 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 1218.20.44112 Boehringer Ingelheim Investigational Site, Ely
  - 1218.20.44101 Boehringer Ingelheim Investigational Site, Guildford
  - 1218.20.44103 Boehringer Ingelheim Investigational Site, Manchester
  - 1218.20.44106 Boehringer Ingelheim Investigational Site, Trowbridge
  - 1218.20.44104 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool
  - 1218.20.44111 Boehringer Ingelheim Investigational Site, Westbury
  - 1218.20.44107 Boehringer Ingelheim Investigational Site, Whitstable

REFERENCES:
- [Derived] Dennis JM, Young KG, Cardoso P, Gudemann LM, McGovern AP, Farmer A, Holman RR, Sattar N, McKinley TJ, Pearson ER, Jones AG, Shields BM, Hattersley AT; MASTERMIND Consortium. A five-drug class model using routinely available clinical features to optimise prescribing in type 2 diabetes: a prediction model development and validation study. Lancet. 2025 Mar 1;405(10480):701-714. doi: 10.1016/S0140-6736(24)02617-5. Epub 2025 Feb 25. PMID 40020703
- [Derived] Gallwitz B, Rosenstock J, Emser A, von Eynatten M, Woerle HJ. Linagliptin is more effective than glimepiride at achieving a composite outcome of target HbA(1)c < 7% with no hypoglycaemia and no weight gain over 2 years. Int J Clin Pract. 2013 Apr;67(4):317-21. doi: 10.1111/ijcp.12101. PMID 23521323
- [Derived] Gallwitz B, Rosenstock J, Rauch T, Bhattacharya S, Patel S, von Eynatten M, Dugi KA, Woerle HJ. 2-year efficacy and safety of linagliptin compared with glimepiride in patients with type 2 diabetes inadequately controlled on metformin: a randomised, double-blind, non-inferiority trial. Lancet. 2012 Aug 4;380(9840):475-83. doi: 10.1016/S0140-6736(12)60691-6. Epub 2012 Jun 28. PMID 22748821
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1218/1218.20_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were in total 1560 patients randomised in the study. Of these, 1 patient was not treated. The remaining 8 patients not accounted for in the treated set were removed from all study analyses (explained in trial report) due to major good-clinical-practice violations at the site, and the inability to verify the validity of any patient level data.
Groups:
- Linagliptin: Patients randomized to receive Linagliptin 5mg and metformin
- Glimepiride: Patients randomized to receive Glimepiride 1-4mg and metformin
Period: Overall Study
Arm/Group | Linagliptin | Glimepiride
Started | 776 (Number who started treatment. One patient in the Linagliptin group was randomized but not treated.) | 775 (Number who started treatment.)
Completed | 587 (Number who completed treatment.) | 604 (Number who completed treatment.)
Not Completed | 189 | 171
Not completed — Lack of Efficacy | 45 | 15
Not completed — Adverse Event | 61 | 90
Not completed — Protocol Violation | 12 | 5
Not completed — Lost to Follow-up | 11 | 13
Not completed — Withdrawal by Subject | 27 | 24
Not completed — Other reason (not specified) | 33 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin | Glimepiride | Total
Number analyzed (Participants) | 776 | 775 | 1551
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (9.4) | 59.8 (9.4) | 59.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 304 | 618
  Male | 462 | 471 | 933
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.21 (4.77) | 30.31 (4.57) | 30.26 (4.67)
Weight [Mean (Standard Deviation); unit: kg] | 86.14 (17.57) | 86.77 (16.69) | 86.46 (17.14)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent] — Baseline HbA1c was available for 1519 patients in the Full Analysis Set (FAS), 764 treated with Linagliptin and 755 patients treated with Glimepiride.
  Percent | 7.69 (0.88) | 7.69 (0.86) | 7.69 (0.87)
Fasting blood plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Baseline fasting plasma glucose (FPG) was available for 1475 patients in the FAS, 740 treated with Linagliptin and 735 patients treated with Glimepiride.
  mg/dL | 164.46 (42.83) | 166.09 (42.05) | 165.27 (42.43)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 52
Description: This co-primary endpoint, change from baseline, reflects the Week 52 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications.
Time Frame: Baseline and week 52
Population: The Full Analysis Set (FAS) included all treated and randomized patients with a baseline and at least one on-treatment HbA1c measurement. Last observation carried forward (LOCF) was used as imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.36 (0.03) | -0.57 (0.03)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Non-Inferiority or Equivalence — The null hypothesis of non-inferiority is rejected if the upper bound of the two-sided 97.5% confidence interval is less than 0.35%. Superiority testing was not part of the pre-specified Week 52 confirmatory analysis; p = 0.0005, ANCOVA — Due to multiple testing of the primary endpoints at weeks 52 and 104 a Bonferroni correction was applied and 97.5% confidence intervals produced. This 1-sided p-value for non-inferiority should be compared to the 1-sided threshold of 0.0125; Least Squares Mean Difference = 0.22, 97.5% CI [0.13 to 0.31], Standard Error of Mean 0.04

2. Primary Outcome: HbA1c Change From Baseline at Week 104
Description: This co-primary endpoint, change from baseline, reflects the Week 104 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications.
Time Frame: Baseline and week 104
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.16 (0.03) | -0.36 (0.03)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Non-Inferiority or Equivalence — The null hypothesis of non-inferiority is rejected if the upper bound of the two-sided 97.5% confidence interval is less than 0.35%. However, superiority testing is only applicable if the Linagliptin decrease is greater than that in Glimepiride; p = 0.0004, ANCOVA — This 1-sided p-value should be compared to the 1-sided threshold of 0.0125 for non-inferiority. Due to the pre-specified hierarchial approach, further confirmatory analysis on the Week24 endpoints is only applicable if superiority is already met; Least Squares Mean Difference = 0.20, 97.5% CI [0.09 to 0.30], Standard Error of Mean 0.05

3. Secondary Outcome: Body Weight Change From Baseline at Week 52
Description: This key secondary endpoint, change from baseline, reflects the Week 52 body weight minus the baseline body weight. Means are treatment adjusted for baseline HbA1c, baseline weight and the number of previous antidiabetic-medications.
Time Frame: Baseline and week 52
Population: This population includes the FAS further restricted to patients with a baseline body weight and one on-treatment body weight measurement. Last observation carried forward (LOCF) was used as imputation rule.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 733 | 722
kg | -1.12 (0.13) | 1.38 (0.14)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p < 0.0001, ANCOVA — This Week52 key secondary endpoint was only to be tested (2-sided threshold of 0.025 to allow for multiple testing within a visit) if the Week52 primary hypothesis was rejected; Least Squares Mean Difference = -2.50, 97.5% CI [-2.91 to -2.09], Standard Error of Mean 0.18

4. Secondary Outcome: Body Weight Change From Baseline at Week 104
Description: This key secondary endpoint, change from baseline, reflects the Week 104 body weight minus the baseline body weight. Means are treatment adjusted for baseline HbA1c, baseline weight and the number of previous antidiabetic-medications.
Time Frame: Baseline and week 104
Population: as for outcome 3
Measure: Mean (Standard Error); unit: kg
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 733 | 722
kg | -1.39 (0.16) | 1.29 (0.16)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p < 0.0001, ANCOVA — Due to testing of multiple endpoints within a visit a sequential testing strategy (at 2-sided threshold of 0.025) was applied to the key secondary endpoints; Least Squares Mean Difference = -2.68, 97.5% CI [-3.17 to -2.19], Standard Error of Mean 0.22

5. Secondary Outcome: Incidence of Hypoglycaemic Events up to 52 Weeks
Description: A hypoglycaemic event is defined as patient showing clinical signs suggestive of low blood glucose confirmed by a home blood glucose monitoring (HBGM) of below 55 mg/dl (3.1 mmol/L)
Time Frame: Week 52
Population: The treated set consisted of all patients treated with at least one dose of study drug
Measure: Number; unit: Patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 776 | 775
Patients | 41 | 249
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — This key secondary endpoint was only to be tested (comparing to a 2-sided threshold of 0.025) if the Week52 body weight change from baseline was confirmatory

6. Secondary Outcome: Incidence of Hypoglycaemic Events up to 104 Weeks
Description: A hypoglycaemic event is defined as patient showing clinical signs suggestive of low blood glucose confirmed by a HBGM of below 55 mg/dl (3.1 mmol/L)
Time Frame: Week 104
Population: The treated set consisted of all patients treated with at least one dose of study drug
Measure: Number; unit: Patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 776 | 775
Patients | 58 | 280
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

7. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at Week 52
Description: This change from baseline reflects the Week 52 FPG minus the Baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and the number of previous anti-diabetic medications.
Time Frame: Baseline and week 52
Population: This population includes the FAS further restricted to patients with a baseline FPG and one on-treatment FPG measurement. Last observation carried forward (LOCF) was used as imputation rule.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 733 | 725
mg/dL | -8.40 (1.25) | -15.24 (1.26)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 6.84, 95% CI [3.51 to 10.16], Standard Error of Mean 1.70

8. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at Week 104
Description: This change from baseline reflects the Week 104 FPG minus the Baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and number of previous anti-diabetic medications.
Time Frame: Baseline and week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 733 | 725
mg/dL | -2.34 (1.46) | -8.72 (1.47)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0012, ANCOVA; Least Squares Mean Difference = 6.38, 95% CI [2.51 to 10.25], Standard Error of Mean 1.97

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 52
Description: The percentage of patients with an HbA1c value below 7.0% at week 52, based upon patients with baseline HbA1c >= 7%. If a patient did not have an HbA1c value at week 52 they were considered a failure, so HbA1c >= 7.0%. The logistic regression is treatment adjusted for baseline HbA1c and number of previous anti-diabetic medications.
Time Frame: Week 52
Population: Full analysis set (FAS) patients with non-completers considered as failures (i.e., non-responders) (NCF) and with baseline HbA1c >=7.0%.
Measure: Number; unit: Percentage of patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 592 | 599
Percentage of patients | 29.6 | 38.9
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; The odds ratio is treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications; Odds Ratio (OR) = 0.625, 95% CI [0.482 to 0.811]

10. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 104
Description: The percentage of patients with an HbA1c value below 7.0% at week 104, based upon patients with baseline HbA1c >= 7%. If a patient did not have an HbA1c value at week 104 they were considered a failure, so HbA1c >= 7.0%. The logistic regression is treatment adjusted for baseline HbA1c and number of previous anti-diabetic medications.
Time Frame: Week 104
Population: as for outcome 9
Measure: Number; unit: Percentage of patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 591 | 593
Percentage of patients | 21.0 | 28.3
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0030, Regression, Logistic; The odds ratio is treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications; Odds Ratio (OR) = 0.654, 95% CI [0.494 to 0.866]

11. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 52
Description: The percentage of patients with an HbA1c value below 6.5% at week 52, based upon patients with baseline HbA1c >= 6.5%. If a patient did not have an HbA1c value at week 52 they were considered a failure, so HbA1c >= 6.5%. The logistic regression is treatment adjusted for baseline HbA1c and number of previous anti-diabetic medications.
Time Frame: Week 52
Population: Full analysis set (FAS) patients with non-completers considered as failures (i.e., non-responders) (NCF) and with baseline HbA1c >=6.5%.
Measure: Number; unit: Percentage of patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 738 | 740
Percentage of patients | 16.9 | 22.7
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0025, Regression, Logistic; The odds ratio is treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications; Odds Ratio (OR) = 0.648, 95% CI [0.489 to 0.859]

12. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 104
Description: The percentage of patients with an HbA1c value below 6.5% at week 104, based upon patients with baseline HbA1c >= 6.5%. If a patient did not have an HbA1c value at week 104 they were considered a failure, so HbA1c >= 6.5%. The logistic regression is treatment adjusted for baseline HbA1c and number of previous anti-diabetic medications.
Time Frame: Week 104
Population: as for outcome 11
Measure: Number; unit: Percentage of patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 736 | 734
Percentage of patients | 10.9 | 14.7
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0240, Regression, Logistic; The odds ratio is treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications; Odds Ratio (OR) = 0.689, 95% CI [0.498 to 0.952]

13. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% at Week 104
Description: Occurrence of relative efficacy response, defined as a lowering of 0.5% HbA1c at week 104
Time Frame: Week 104
Population: FAS (NCF)
Measure: Number; unit: Percentage of patients
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percentage of patients | 26.2 | 33.5
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; The odds ratio is treatment adjusted for baseline HbA1c and the number of previous anti-diabetic medications; Odds Ratio (OR) = 0.700, 95% CI [0.560 to 0.875]

14. Secondary Outcome: 2 hr Postprandial Glucose (PPG) Change From Baseline at Week 104
Description: This change from baseline reflects the Week 104 2 hr PPG minus the Baseline 2hr PPG. Means are treatment adjusted for baseline HbA1c, baseline 2hr PPG and number of previous anti-diabetic medications.
Time Frame: Baseline and week 104
Population: Patients in the FAS with a valid meal tolerance test (MTT) at baseline and at least one valid on-treatment MTT (MTT104).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 212 | 222
mg/dL | -28.47 (4.32) | -18.72 (4.28)
Statistical Analysis 1: Comparison: Linagliptin vs Glimepiride; Linagliptin versus Glimepiride; Test type: Superiority or Other; p = 0.0918, ANCOVA; Least Squares Mean Difference = -9.47, 95% CI [-21.07 to 1.59], Standard Error of Mean 5.77

15. Secondary Outcome: HbA1c Change at Week 4
Description: Difference of base percent value [Week x(%) - baseline (%)]
Time Frame: Baseline and week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.26 (0.41) | -0.33 (0.46)

16. Secondary Outcome: HbA1c Change at Week 8
Time Frame: Baseline and week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.37 (0.59) | -0.58 (0.62)

17. Secondary Outcome: HbA1c Change at Week 12
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.43 (0.64) | -0.75 (0.69)

18. Secondary Outcome: HbA1c Change at Week 16
Time Frame: Baseline and week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.45 (0.66) | -0.78 (0.73)

19. Secondary Outcome: HbA1c Change at Week 28
Time Frame: Baseline and week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.43 (0.73) | -0.74 (0.81)

20. Secondary Outcome: HbA1c Change at Week 40
Time Frame: Baseline and week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.42 (0.77) | -0.69 (0.83)

21. Secondary Outcome: HbA1c Change at Week 52
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.41 (0.82) | -0.63 (0.85)

22. Secondary Outcome: HbA1c Change at Week 65
Time Frame: Baseline and week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.32 (0.91) | -0.53 (0.87)

23. Secondary Outcome: HbA1c Change at Week 78
Time Frame: Baseline and week 78
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.22 (0.92) | -0.43 (0.90)

24. Secondary Outcome: HbA1c Change at Week 91
Time Frame: Baseline and week 91
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.21 (0.94) | -0.43 (0.90)

25. Secondary Outcome: HbA1c Change at Week 104
Description: The Full Analysis Set (FAS) included all treated and randomized patients with a baseline and at least one on-treatment HbA1c measurement available during the first phase of the study. Last observation carried forward (LOCF) was used as imputation rule.
Time Frame: Baseline and week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 764 | 755
Percent | -0.21 (0.95) | -0.41 (0.93)

26. Secondary Outcome: Change in Baseline Lipid Parameter Cholesterol at Week 104
Time Frame: Baseline and week 104
Population: This population includes the treated set (all patients treated with at least one dose of study drug), and non-missing laboratory data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 741 | 726
mg/dL | 0 (14) | 1 (14)

27. Secondary Outcome: Change in Baseline Lipid Parameter HDL at Week 104
Time Frame: Baseline and week 104
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 740 | 725
mg/dl | 1 (9) | 0 (9)

28. Secondary Outcome: Change in Baseline Lipid Parameter Low Density Lipoprotein (LDL) at Week 104
Time Frame: Baseline and week 104
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 734 | 720
mg/dL | 1 (23) | 3 (25)

29. Secondary Outcome: Change in Baseline Lipid Parameter Triglyceride at Week 104
Time Frame: Baseline and week 104
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Linagliptin | Glimepiride
Number analyzed (Participants) | 740 | 725
mg/dL | -11 (153) | -7 (148)

ADVERSE EVENTS:
Time Frame: From day of first dose until 7 days after last dose
Arm/Group | Linagliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 135/776 | 162/775
Other Adverse Events (participants affected / at risk) | 438/776 | 526/775
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin (N=776) | Glimepiride (N=775)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 4
Angina pectoris (Cardiac disorders) | 5 | 4
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 3 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 5 | 6
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve disease mixed (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 6
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 0
Central nervous system dermoid tumour (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Goitre (Endocrine disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 1 | 1
Optic disc haemorrhage (Eye disorders) | 0 | 1
Optic neuropathy (Eye disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Drowning (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mass (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 3 | 3
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Balanitis candida (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 3
Erysipelas (Infections and infestations) | 2 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 4
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 3
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Accident (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 3 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 6
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Agnosia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 4
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 6
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 5
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium tremens (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Paranoia (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Renal colic (Renal and urinary disorders) | 1 | 4
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Penile curvature (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin (N=776) | Glimepiride (N=775)
Diarrhoea (Gastrointestinal disorders) | 52 | 60
Nausea (Gastrointestinal disorders) | 37 | 39
Bronchitis (Infections and infestations) | 50 | 60
Nasopharyngitis (Infections and infestations) | 124 | 125
Upper respiratory tract infection (Infections and infestations) | 62 | 59
Urinary tract infection (Infections and infestations) | 49 | 51
Hyperglycaemia (Metabolism and nutrition disorders) | 39 | 40
Hypoglycaemia (Metabolism and nutrition disorders) | 55 | 267
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 68 | 65
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 | 30
Dizziness (Nervous system disorders) | 26 | 47
Headache (Nervous system disorders) | 50 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 38
Hypertension (Vascular disorders) | 48 | 60

LIMITATIONS AND CAVEATS:
With the exception of HbA1c<6.5% and HbA1c<7.0% at Week52, all other endpoints are presented in the Week52 repeated analysis within the final clinical trial report, where discrepancies between interim and final results are also explained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.